CLINICAL TRIAL: NCT03044457
Title: Forgotten Joint Score After Reversed Gap Technique vs. Gap Technique
Brief Title: Forgotten Joint Score After Reversed Gap Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Georg Matziolis, Director of the Orthopaedic Department, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCAFJS
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Total Knee Arthroplasty; Clinical Outcome

STUDY DESIGN:
Intervention Model Description: Two groups: "reversed gap technique" vs. "gap technique", randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: neither the participant nor the outcome assessor know the group. The surgeon of course knows.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TKA by reversed gap technique (Experimental): new operative technique of positioning the femoral and tibial component based on soft tissue tension and femoral 3D geometry.
  Interventions: Procedure: TKA
- TKA by gap technique (Active Comparator): standard operative technique serving as control. tibia component positioning according to the mechanical axis, femoral component positioning according to the mechanical axis and soft tissue tension in flexion
  Interventions: Procedure: TKA

INTERVENTIONS:
Procedure: TKA — femoral and tibial positioning using the "reversed gap technique"

SUMMARY:
A new operation technique was established ("reversed gap technique" for implantation of total knee arthroplasties. Based on the encouraging results of a pilot study, the clinical outcome shall be evaluated using the conventional "gap technique" as control in a RCT study.

ELIGIBILITY:
Inclusion Criteria:

* indication for implantation a total knee arthroplasty

Exclusion Criteria:

* indication for a constrained implant
* secondary type of arthritis (rheumatoid, post traumatic, post infectious)
* former "open" surgery on the joint using an arthrotomy or HTO (arthroscopy excluded)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score 12 | one year after operation
  clinical score

IPD SHARING:
Plan to Share IPD: No